CLINICAL TRIAL: NCT01341782
Title: Comparison of Efficacy and Safety of Paricalcitol Injection With Maxacalcitol Injection in Adult Japanese Chronic Kidney Disease Subjects Receiving Hemodialysis With Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M11-517
Record Dates: First submitted 2011-04-25; First posted 2011-04-26 (Estimated); Results first posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-04

CONDITIONS: Secondary Hyperparathyroidism; Hemodialysis
Keywords: Secondary hyperparathyroidism; Paricalcitol; Hemodialysis; Maxacalcitol
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — paricalcitol; maxacalcitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paricalcitol (Experimental): Participants received paricalcitol at an initial dose of 2 µg, and maxacalcitol placebo administered 3 times per week at each hemodialysis via intravenous catheter for 12 weeks. After 2 weeks the dose could be adjusted ± 1 µg based on protocol-specified criteria up to a maximum of 7 µg.
  Interventions: Drug: paricalcitol; Drug: maxacalcitol placebo
- Maxacalcitol (Active Comparator): Participants received maxacalcitol at an initial dose of 5 µg (iPTH < 500 pg/mL at Screening) or 10 µg (iPTH ≥ 500 pg/mL at Screening), and paricalcitol placebo administered 3 times per week at each hemodialysis via intravenous catheter for 12 weeks. After 2 weeks the dose could be adjusted ± 2.5 µg based on protocol-specified criteria up to a maximum of 20 µg.
  Interventions: Drug: maxacalcitol; Drug: paricalcitol placebo

INTERVENTIONS:
Drug: paricalcitol
  Other Names: ABT-358; Zemplar
  Arms: Paricalcitol
Drug: maxacalcitol
  Other Names: oxarol
  Arms: Maxacalcitol
Drug: paricalcitol placebo
  Arms: Maxacalcitol
Drug: maxacalcitol placebo
  Arms: Paricalcitol

SUMMARY:
This study is a comparison of the efficacy and safety of paricalcitol injection with maxacalcitol injection in adult Japanese chronic kidney disease patients receiving hemodialysis with secondary hyperparathyroidism. The main objective of this study is to demonstrate the efficacy of paricalcitol injection in reducing levels of parathyroid hormone without clinically significant hypercalcemia, compared to maxacalcitol injection.

ELIGIBILITY:
Inclusion Criteria:

* Adult Chronic Kidney Disease (CKD) Stage 5 patients undergoing dialysis with stable dialysate calcium and phosphate binders
* On three times weekly hemodialysis for at least 3 months prior with intact parathyroid hormone (iPTH) greater than or equal to 300 pg/mL, adjusted normalized serum total calcium (Ca) greater than or equal to 8.4 to less than 10.2 mg/dL, serum phosphorus (P) less than or equal to 6.5 mg/dL.

Exclusion Criteria:

* Patients with a recent history of severe cardiovascular or hepatic disease, uncontrolled hypertension or uncontrolled diabetes
* Patients who have received a parathyroidectomy or ethanol infusion within the prior year
* Patients taking drugs that affect iPTH, calcium or bone metabolism
* Patients who will need to take chronic doses (greater than or equal to 2 consecutive weeks) of cytochrome P450 inhibitors (e.g., clarithromycin, grapefruit products) or inducers (e.g., carbamazepine, rifampicin)
* Female patients who are pregnant, possibly pregnant, wish to become pregnant, or participate in breastfeeding during the study period.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuya Kobayashi, BA, Study Director — AbbVie
Locations (45):
- Japan (45):
  - Site Reference ID/Investigator# 53485, Aichi
  - Site Reference ID/Investigator# 51571, Chiba
  - Site Reference ID/Investigator# 52963, Chiba
  - Site Reference ID/Investigator# 52966, Chiba
  - Site Reference ID/Investigator# 51578, Gifu
  - Site Reference ID/Investigator# 52965, Gunma
  - Site Reference ID/Investigator# 53782, Hadano
  - Site Reference ID/Investigator# 57483, Himeji
  - Site Reference ID/Investigator# 57487, Hokkaido
  - Site Reference ID/Investigator# 53484, Hyōgo
  - Site Reference ID/Investigator# 54385, Ibaraki
  - Site Reference ID/Investigator# 51581, Kagawa
  - Site Reference ID/Investigator# 59164, Kagoshima
  - Site Reference ID/Investigator# 51574, Kanagawa
  - Site Reference ID/Investigator# 51575, Kanagawa
  - Site Reference ID/Investigator# 52751, Kodaira
  - Site Reference ID/Investigator# 62025, Koga
  - Site Reference ID/Investigator# 54384, Matsumoto
  - Site Reference ID/Investigator# 52745, Midori
  - Site Reference ID/Investigator# 51569, Mito
  - Site Reference ID/Investigator# 52964, Nagano
  - Site Reference ID/Investigator# 53483, Nagano
  - Site Reference ID/Investigator# 51582, Nagasaki
  - Site Reference ID/Investigator# 54388, Nagoya
  - Site Reference ID/Investigator# 51576, Niigata
  - Site Reference ID/Investigator# 51577, Niigata
  - Site Reference ID/Investigator# 51580, Osaka
  - Site Reference ID/Investigator# 52747, Osaka
  - Site Reference ID/Investigator# 52748, Osaka
  - Site Reference ID/Investigator# 52750, Osaka
  - Site Reference ID/Investigator# 51570, Saitama
  - Site Reference ID/Investigator# 54387, Sakai
  - Site Reference ID/Investigator# 52746, Sapporo
  - Site Reference ID/Investigator# 51579, Shizuoka
  - Site Reference ID/Investigator# 62024, Takasaki
  - Site Reference ID/Investigator# 51572, Tokyo
  - Site Reference ID/Investigator# 52752, Tokyo
  - Site Reference ID/Investigator# 53482, Tokyo
  - Site Reference ID/Investigator# 59162, Tokyo
  - Site Reference ID/Investigator# 59966, Tokyo
  - Site Reference ID/Investigator# 53783, Tomakomai-shi
  - Site Reference ID/Investigator# 54383, Toyama
  - Site Reference ID/Investigator# 52749, Wakayama
  - Site Reference ID/Investigator# 52962, Yachiyoshi
  - Site Reference ID/Investigator# 59163, Yokohama

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Maxacalcitol: Participants received maxacalcitol at an initial dose of 5 µg (intact parathyroid hormone [iPTH] < 500 pg/mL at Screening) or 10 µg (iPTH ≥ 500 pg/mL at Screening), and paricalcitol placebo administered 3 times per week at each hemodialysis via intravenous catheter for 12 weeks. After 2 weeks the dose could be adjusted ± 2.5 µg based on protocol-specified criteria up to a maximum of 20 µg.
Period: Overall Study
Arm/Group | Paricalcitol | Maxacalcitol
Started | 127 | 128
Completed | 112 | 114
Not Completed | 15 | 14
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Missed 3 consecutive doses | 0 | 4
Not completed — 2 consecutive calcium values >11.5 mg/dL | 0 | 1
Not completed — 2 consecutive calcium values < 8.4 mg/dL | 3 | 3
Not completed — Other | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paricalcitol | Maxacalcitol | Total
Number analyzed (Participants) | 127 | 128 | 255
Age Continuous [Mean (Standard Deviation); unit: years] | 61.5 (11.24) | 61.6 (12.46) | 61.6 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 47 | 92
  Male | 82 | 81 | 163
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 127 | 128 | 255
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 127 | 128 | 255
Duration of hemodialysis [Mean (Standard Deviation); unit: years] | 8.4 (6.73) | 8.9 (7.50) | 8.6 (7.12)
Intact parathyroid hormone level [Mean (Standard Deviation); unit: pg/mL] | 525.4 (205.55) | 527.1 (203.33) | 526.3 (204.03)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Target Intact Parathyroid Hormone (iPTH) and Without Hypercalcemia
Description: The target iPTH range was 60-180 pg/mL, based on the average of the last 3 weeks of treatment, and with no hypercalcemia during the treatment phase. Hypercalcemia was defined as at least 1 corrected calcium value > 11.0 mg/dL or at least 2 corrected calcium values ≥ 10.5 mg/dL. iPTH was measured before the first dialysis session of each week and analyzed by the central laboratory.
Time Frame: iPTH measured during the last three weeks of treatment (Weeks 11, 12, and 13). Calcium measured throughout the study (Weeks 1-13).
Population: The per-protocol set (PPS) consists of all randomized patients who completed at least 8 weeks of treatment and met the conditions specified by the subject classification (i.e., no violation of inclusion/exclusion criteria) that occurred before the study blind was broken.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paricalcitol | Maxacalcitol
Number analyzed (Participants) | 119 | 118
percentage of participants | 27.7 [19.92 to 36.68] | 30.5 [22.37 to 39.66]

2. Secondary Outcome: Percentage of Participants With ≥ 50% Reduction in Intact Parathyroid Hormone (iPTH) From Baseline and With No Hypercalcemia
Description: The percentage of participants with greater than or equal to 50% reduction in intact parathyroid hormone (iPTH) from baseline to the average of the last 3 weeks of treatment and with no hypercalcemia during the treatment phase. iPTH was measured before the first dialysis session of each week and analyzed by the central laboratory. Hypercalcemia was defined as at least 1 corrected calcium value > 11.0 mg/dL or at least 2 corrected calcium values ≥ 10.5 mg/dL.
Time Frame: Baseline to the last three weeks of treatment (Weeks 11, 12, and 13) for iPTH. Calcium measured throughout the study (Weeks 1-13).
Population: The Full Analysis Set (FAS) consists of all randomized patients who received at least 1 dose of study drug and had at least 1 post-baseline iPTH measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paricalcitol | Maxacalcitol
Number analyzed (Participants) | 127 | 128
percentage of participants | 34.6 [26.43 to 43.60] | 39.1 [30.56 to 48.08]

3. Secondary Outcome: Percentage of Participants With Target Intact Parathyroid Hormone (iPTH)
Description: The target iPTH range was 60-180 pg/mL, based on the average of the last 3 weeks of treatment. iPTH was measured before the first dialysis session of each week and analyzed by the central laboratory.
Time Frame: The last three weeks of treatment (Weeks 11, 12, and 13)
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paricalcitol | Maxacalcitol
Number analyzed (Participants) | 127 | 128
percentage of participants | 31.5 [23.55 to 40.33] | 32.8 [24.78 to 41.67]

4. Secondary Outcome: Percentage of Participants With ≥ 50% Reduction in Intact Parathyroid Hormone (iPTH) From Baseline
Description: The percentage of participants with a greater than or equal to 50% reduction in intact parathyroid hormone (iPTH) from baseline to the average of the last 3 weeks of treatment. iPTH was measured before the first dialysis session of each week and analyzed by the central laboratory.
Time Frame: Baseline to the last three weeks of treatment (Weeks 11, 12, and 13)
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paricalcitol | Maxacalcitol
Number analyzed (Participants) | 127 | 128
percentage of participants | 44.9 [36.05 to 53.96] | 50.8 [41.80 to 59.72]

5. Secondary Outcome: Number of Visits at Which Participants Achieved iPTH Control With ≥ 50% Reduction in Intact Parathyroid Hormone (iPTH) From Baseline
Description: iPTH control was defined as a ≥ 50% reduction from baseline. iPTH was measured before the first dialysis session of the week, each week during the treatment phase and analyzed by the central laboratory.
Time Frame: Weeks 2 to 13
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Paricalcitol | Maxacalcitol
Number analyzed (Participants) | 127 | 128
visits | 3.9 (2.97) | 5.3 (3.17)

6. Secondary Outcome: Number of Visits at Which Participants Achieved iPTH Control in the Target Range of 60 to 180 pg/mL
Description: iPTH control was defined as being within the target range of 60 to 180 pg/mL. iPTH was measured before the first dialysis session of the week, once a week during the treatment phase and analyzed by the central laboratory.
Time Frame: Weeks 2 to 13
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Paricalcitol | Maxacalcitol
Number analyzed (Participants) | 127 | 128
visits | 2.6 (2.51) | 3.4 (2.84)

ADVERSE EVENTS:
Arm/Group | Paricalcitol | Maxacalcitol
Serious Adverse Events (participants affected / at risk) | 10/127 | 15/128
Other Adverse Events (participants affected / at risk) | 118/127 | 123/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol (N=127) | Maxacalcitol (N=128)
Myocardial infarction (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Parathyroid gland enlargement (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 0 | 2
Shunt stenosis (Injury, poisoning and procedural complications) | 2 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Thalamus haemorrhage (Nervous system disorders) | 1 | 0
Renal disorder in pregnancy (Renal and urinary disorders) | 0 | 1 — The patient was not pregnant during the study, but had a past medical history of pregnancy-induced kidney disorder
Prostatitis (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol (N=127) | Maxacalcitol (N=128)
Constipation (Gastrointestinal disorders) | 10 | 7
Diarrhoea (Gastrointestinal disorders) | 11 | 6
Vomiting (Gastrointestinal disorders) | 11 | 7
Nasopharyngitis (Infections and infestations) | 43 | 49
Contusion (Injury, poisoning and procedural complications) | 8 | 7
Excoriation (Injury, poisoning and procedural complications) | 9 | 2 — All excoriation events in this study were trauma-related
Procedural hypotension (Injury, poisoning and procedural complications) | 14 | 20
Shunt stenosis (Injury, poisoning and procedural complications) | 9 | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 50 | 55
Hyperphosphataemia (Metabolism and nutrition disorders) | 21 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 6
Hypertension (Vascular disorders) | 20 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.